CLINICAL TRIAL: NCT03071302
Title: Evaluation of Tomographic and Genetic Aspects of Keratoconus Patients Compared to Sounds Corneas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Gildasio Castello de Almeida Junior, PROF. DR., Sao Jose do Rio Preto Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CAAE 44071315.7.0000.5415; 2015/17226-7 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2017-02-28; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Keratoconus; Keratoconus, Unspecified, Bilateral
Keywords: Keratoconus,Corneal Dystrophies, corneal Tomography, topography
MeSH Terms: conditions — Keratoconus; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- keratoconus (Active Comparator): Evaluation of Visual System Homeobox 1 (VSX1), Superoxide Dismutase (SOD1), Tissue Inhibitors of Metalloproteinases (TIMP3) genes. Keratoconus with fellow eye without topographic and tomographic keratoconous pattern.Evaluation of tomographic datas. Sometimes we picked up the sample of corneal epithelium, and peripheral blood sample from corneal cross linking surgeries, in that case of keratoconus progression.
  Group A Keratoconus/ like sound cornea. Group C Keratoconus / Keratoconus
  Group C Keratoconus / Keratoconus
  Interventions: Other: EVALUATION OF VSX1, SOD1, and TIMP3 genes
- sound cornea (Placebo Comparator): Evaluation of VSX1, SOD1, and TIMP3 genes. To analyze tomographic aspects, we evaluated the patients that underwent to LASIK (Lasei in situ Keratomileusis) with 2 year with follow up without any sign of ectasia To analyze the genes we picked up the sample of corneal epithelium, and peripheral blood sample from PRK (PhotoRefractive Keratectomy) surgeries. These patients showed topographic and tomographic normal pattern.
  Group B Sound Cornea / Sound Cornea
  Interventions: Other: EVALUATION OF VSX1, SOD1, and TIMP3 genes

INTERVENTIONS:
Other: EVALUATION OF VSX1, SOD1, and TIMP3 genes — Evaluation of VISX1, SOD1, TIMP3 genes in corneal epithelium, and in peripheral blood. Evaluation of pentacam parameters
  Other Names: pentacam and gene evaluation

SUMMARY:
Evaluation of tomographic (Pentacam) parameters and genetic parameters of Visual System Homeobox 1 (VSX1), Superoxide Dismutase (SOD1), Tissue Inhibitors of Metalloproteinases (TIMP3) genes of keratoconus patients diagnosed by clinical exam and topographic pattern. Basically we are screening patients that don't have keratoconus that those have keratoconus. The pentacam index of corneal curvature, thinnest point, corneal high order aberrations, posterior and anterior elevation, corneal densitometry, corneal volume were investigated. To analyze the genes, we took corneal epithelium samples of patients submitted to cross linking compared to (PRK) Photo Refractive Keratectomy ones. Also will be evaluated the genes of peripheral blood.

DETAILED DESCRIPTION:
Keratoconus is a common disease that affects the cornea in both genders in all ethnic groups and that can manifest unilaterally or bilaterally in patients. Keratoconus due to a degenerative disease, its progression can be fast in various situations, affecting 1 in every 2,000 people, what results in severe structural changes of the cornea, which reduces its thickness and modify its normal curvature to a more conical shape. Keratoconus arises in adolescence and lasts for thirty to forty years of age, where it stabilizes and it is considered a major cause of corneal transplantation. Factors such as atopy, overuse of contact lenses and the act of rubbing the eyes are also related to the disease. The clinical picture consists of a lot of varied symptoms and it depends on the stage of disease progression. Currently it is known that genetic and environmental factors are involved in the desease emergence. Recently several genetic studies have aimed to identify mutations in genes which are directly linked to Keratoconus, such as VSX1, SOD1 and TIMP3 genes. However, despite the efforts directed towards the understanding of the genetic aspects of this disease, involving many genes, there are still many questions about the role of these genes in Keratoconus etiology. Thus, the present study aims to identify the presence of mutations in VSX1, SOD1 and TIMP3 genes, which are considered important candidates for the origin and development of this eye anomaly, through the analysis of their nucleotide sequences in corneal tissue and peripheral blood in Keratoconus patients, in their unilateral and bilateral forms. The results will allow to compare the presented mutations in different analysed tissues for unilateral and bilateral forms of Keratoconus and also compare them with the same tissues in healthy patients, in an attempt to establish what the likely inherited and/or acquired genetic mutations are causing this condition. Thus providing genetic data, still unpublished in Brazilian populations, which may offer subsidies for the characterization of the mutation dynamics and their patterns, on the origin and development of Keratoconus. Also will be evaluated the tomographic index as corneal curvature, thinnest point, corneal high order aberrations, posterior and anterior elevation, corneal densitometry, corneal volume. The idea is focused on that suspicious cornea that has the fellow eye with unequivocal keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with keratoconus in clinical examination, topography and tomography
* Patients with clinical examination, topography, and tomography aspect of sound cornea in one eye, and the fellow eye diagnosed with keratoconus by clinical examination, topography, and tomography.

Patients diagnosed with keratoconus by clinical examination, topography, and tomography in both eyes (OU).

* Patients with some degree of ametropia that underwent to PRK and LASIK

Exclusion Criteria:

* History of eye trauma, glaucoma, dysfunctional tear syndrome, rosacea, neurotrophic keratopathy, systemic or topical use of immunosuppressive drugs, previous ocular surgeries.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 210 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the tomographic parameters of keratoconus, subclinical keratoconus in relation to sound corneas and identify the mutations present in the genes VSX1, SOD1 and TIMP3 in individuals affected by keratoconus. | 18 months
  The aim of this study was to evaluate Evaluate the tomographic parameters of keratoconus, subclinical keratoconus in relation to sound corneas and identify the mutations present in the genes VSX1, SOD1 and TIMP3 in individuals affected by keratoconus in several forms of manifestation.

SECONDARY OUTCOMES:
Tomographic parameters | 18 months
  Evaluating whether cross-referencing of known indexes may improve sensitivity and specificity in the detection of subclinical keratoconus;
  - Evaluate if there is a correlation between the different tomographic indices; To evaluate the cornea densitometry in patients with keratoconus and its absence.
Genetic evaluation, VISX1, SOD1, TIMP3 | 18 months
  Avalue if after removal of the epithelium there is a very large change in the curvature, elevations and topometry of the cornea;
  * Identify the presence of mutations in the VSX1, SOD1 and TIMP3 genes, from nucleotide sequence analysis in tissues of the affected cornea, normal cornea and peripheral blood, in patients with this pathology in their several forms.
  * Compare the mutations present in the different tissues analyzed, for the unilateral and bilateral forms of keratoconus and also to compare them with the same tissues in healthy patients;
  * Establish which are the probable inherited and / or acquired genetic mutations that cause this pathology, from the analysis of the same in the peripheral blood of the affected individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio C Almeida Jr, MD, PhD, Principal Investigator — FAMERP, Visum Eye Center
Locations (1):
- Visum Eye Center / Immunogenetic laboratory of FAMERP, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bisceglia L, De Bonis P, Pizzicoli C, Fischetti L, Laborante A, Di Perna M, Giuliani F, Delle Noci N, Buzzonetti L, Zelante L. Linkage analysis in keratoconus: replication of locus 5q21.2 and identification of other suggestive Loci. Invest Ophthalmol Vis Sci. 2009 Mar;50(3):1081-6. doi: 10.1167/iovs.08-2382. Epub 2008 Oct 31. PMID 18978346
- [Background] Karolak JA, Gajecka M. Genomic strategies to understand causes of keratoconus. Mol Genet Genomics. 2017 Apr;292(2):251-269. doi: 10.1007/s00438-016-1283-z. Epub 2016 Dec 28. PMID 28032277
- [Result] Li X, Yang H, Rabinowitz YS. Longitudinal study of keratoconus progression. Exp Eye Res. 2007 Oct;85(4):502-7. doi: 10.1016/j.exer.2007.06.016. Epub 2007 Jul 6. PMID 17681291
- [Result] Abu-Amero KK, Kalantan H, Al-Muammar AM. Analysis of the VSX1 gene in keratoconus patients from Saudi Arabia. Mol Vis. 2011 Mar 8;17:667-72. PMID 21403853
- [Result] Alio JL, Shabayek MH. Corneal higher order aberrations: a method to grade keratoconus. J Refract Surg. 2006 Jun;22(6):539-45. doi: 10.3928/1081-597X-20060601-05. PMID 16805116
- [Result] Ambrosio R Jr, Alonso RS, Luz A, Coca Velarde LG. Corneal-thickness spatial profile and corneal-volume distribution: tomographic indices to detect keratoconus. J Cataract Refract Surg. 2006 Nov;32(11):1851-9. doi: 10.1016/j.jcrs.2006.06.025. PMID 17081868
- [Result] Ambrosio R Jr, Caiado AL, Guerra FP, Louzada R, Sinha RA, Luz A, Dupps WJ, Belin MW. Novel pachymetric parameters based on corneal tomography for diagnosing keratoconus. J Refract Surg. 2011 Oct;27(10):753-8. doi: 10.3928/1081597X-20110721-01. Epub 2011 Jul 29. PMID 21800785
- [Result] Arnal E, Peris-Martinez C, Menezo JL, Johnsen-Soriano S, Romero FJ. Oxidative stress in keratoconus? Invest Ophthalmol Vis Sci. 2011 Nov 4;52(12):8592-7. doi: 10.1167/iovs.11-7732. PMID 21969298
- [Result] Bae GH, Kim JR, Kim CH, Lim DH, Chung ES, Chung TY. Corneal topographic and tomographic analysis of fellow eyes in unilateral keratoconus patients using Pentacam. Am J Ophthalmol. 2014 Jan;157(1):103-109.e1. doi: 10.1016/j.ajo.2013.08.014. Epub 2013 Oct 25. PMID 24452012
- [Result] Beckh U, Schonherr U, Naumann GO. [Autosomal dominant keratoconus as the chief ocular symptom in Lobstein osteogenesis imperfecta tarda]. Klin Monbl Augenheilkd. 1995 Apr;206(4):268-72. doi: 10.1055/s-2008-1035438. German. PMID 7791289
- [Result] Behndig A, Karlsson K, Johansson BO, Brannstrom T, Marklund SL. Superoxide dismutase isoenzymes in the normal and diseased human cornea. Invest Ophthalmol Vis Sci. 2001 Sep;42(10):2293-6. PMID 11527942
- [Result] Bardak H, Gunay M, Yildiz E, Bardak Y, Gunay B, Ozbas H, Bagci O. Novel visual system homeobox 1 gene mutations in Turkish patients with keratoconus. Genet Mol Res. 2016 Nov 3;15(4). doi: 10.4238/gmr15049024. PMID 27819732
- [Result] Bykhovskaya Y, Margines B, Rabinowitz YS. Genetics in Keratoconus: where are we? Eye Vis (Lond). 2016 Jun 27;3:16. doi: 10.1186/s40662-016-0047-5. eCollection 2016. PMID 27350955
- [Result] Chen D, Lam AK. Intrasession and intersession repeatability of the Pentacam system on posterior corneal assessment in the normal human eye. J Cataract Refract Surg. 2007 Mar;33(3):448-54. doi: 10.1016/j.jcrs.2006.11.008. PMID 17321396
- [Result] Chow RL, Volgyi B, Szilard RK, Ng D, McKerlie C, Bloomfield SA, Birch DG, McInnes RR. Control of late off-center cone bipolar cell differentiation and visual signaling by the homeobox gene Vsx1. Proc Natl Acad Sci U S A. 2004 Feb 10;101(6):1754-9. doi: 10.1073/pnas.0306520101. Epub 2004 Jan 26. PMID 14745032
- [Result] Collier SA. Is the corneal degradation in keratoconus caused by matrix-metalloproteinases? Clin Exp Ophthalmol. 2001 Dec;29(6):340-4. doi: 10.1046/j.1442-9071.2001.d01-17.x. PMID 11778801
- [Result] Galvis V, Sherwin T, Tello A, Merayo J, Barrera R, Acera A. Keratoconus: an inflammatory disorder? Eye (Lond). 2015 Jul;29(7):843-59. doi: 10.1038/eye.2015.63. Epub 2015 May 1. PMID 25931166
- [Result] Sugar J, Macsai MS. What causes keratoconus? Cornea. 2012 Jun;31(6):716-9. doi: 10.1097/ICO.0b013e31823f8c72. PMID 22406940
- [Result] Kenney MC, Brown DJ, Rajeev B. Everett Kinsey lecture. The elusive causes of keratoconus: a working hypothesis. CLAO J. 2000 Jan;26(1):10-3. PMID 10656302
- [Result] De Bonis P, Laborante A, Pizzicoli C, Stallone R, Barbano R, Longo C, Mazzilli E, Zelante L, Bisceglia L. Mutational screening of VSX1, SPARC, SOD1, LOX, and TIMP3 in keratoconus. Mol Vis. 2011;17:2482-94. Epub 2011 Sep 24. PMID 21976959
- [Result] Driver PJ, Reed JW, Davis RM. Familial cases of keratoconus associated with posterior polymorphous dystrophy. Am J Ophthalmol. 1994 Aug 15;118(2):256-7. doi: 10.1016/s0002-9394(14)72911-3. No abstract available. PMID 8053477
- [Result] Edwards M, McGhee CN, Dean S. The genetics of keratoconus. Clin Exp Ophthalmol. 2001 Dec;29(6):345-51. doi: 10.1046/j.1442-9071.2001.d01-16.x. PMID 11778802
- [Result] Greenstein SA, Fry KL, Bhatt J, Hersh PS. Natural history of corneal haze after collagen crosslinking for keratoconus and corneal ectasia: Scheimpflug and biomicroscopic analysis. J Cataract Refract Surg. 2010 Dec;36(12):2105-14. doi: 10.1016/j.jcrs.2010.06.067. PMID 21111314
- [Result] Grzybowski A, McGhee CN. The early history of keratoconus prior to Nottingham's landmark 1854 treatise on conical cornea: a review. Clin Exp Optom. 2013 Mar;96(2):140-5. doi: 10.1111/cxo.12035. Epub 2013 Feb 18. PMID 23414219
- [Result] Gunes A, Tok L, Tok O, Seyrek L. The Youngest Patient with Bilateral Keratoconus Secondary to Chronic Persistent Eye Rubbing. Semin Ophthalmol. 2015;30(5-6):454-6. doi: 10.3109/08820538.2013.874480. Epub 2014 Feb 7. PMID 24506444
- [Result] Heon E, Greenberg A, Kopp KK, Rootman D, Vincent AL, Billingsley G, Priston M, Dorval KM, Chow RL, McInnes RR, Heathcote G, Westall C, Sutphin JE, Semina E, Bremner R, Stone EM. VSX1: a gene for posterior polymorphous dystrophy and keratoconus. Hum Mol Genet. 2002 May 1;11(9):1029-36. doi: 10.1093/hmg/11.9.1029. PMID 11978762
- [Result] Heon E, Mathers WD, Alward WL, Weisenthal RW, Sunden SL, Fishbaugh JA, Taylor CM, Krachmer JH, Sheffield VC, Stone EM. Linkage of posterior polymorphous corneal dystrophy to 20q11. Hum Mol Genet. 1995 Mar;4(3):485-8. doi: 10.1093/hmg/4.3.485. PMID 7795607
- [Result] Hirano M, Hung WY, Cole N, Azim AC, Deng HX, Siddique T. Multiple transcripts of the human Cu,Zn superoxide dismutase gene. Biochem Biophys Res Commun. 2000 Sep 16;276(1):52-6. doi: 10.1006/bbrc.2000.3427. PMID 11006081
- [Result] Hughes AE, Dash DP, Jackson AJ, Frazer DG, Silvestri G. Familial keratoconus with cataract: linkage to the long arm of chromosome 15 and exclusion of candidate genes. Invest Ophthalmol Vis Sci. 2003 Dec;44(12):5063-6. doi: 10.1167/iovs.03-0399. PMID 14638698
- [Result] Ishii R, Kamiya K, Igarashi A, Shimizu K, Utsumi Y, Kumanomido T. Correlation of corneal elevation with severity of keratoconus by means of anterior and posterior topographic analysis. Cornea. 2012 Mar;31(3):253-8. doi: 10.1097/ICO.0B013E31823D1EE0. PMID 22316650
- [Result] Jeoung JW, Kim MK, Park SS, Kim SY, Ko HS, Wee WR, Lee JH. VSX1 gene and keratoconus: genetic analysis in Korean patients. Cornea. 2012 Jul;31(7):746-50. doi: 10.1097/ICO.0b013e3181e16dd0. PMID 22531431
- [Result] Mok JW, Baek SJ, Joo CK. VSX1 gene variants are associated with keratoconus in unrelated Korean patients. J Hum Genet. 2008;53(9):842-849. doi: 10.1007/s10038-008-0319-6. Epub 2008 Jul 15. PMID 18626569
- [Result] Akcay EK, Uysal BS, Sarac O, Ugurlu N, Yulek F, Cagil N, Aslan N. The Effect of Corneal Epithelium on Corneal Curvature in Patients with Keratoconus. Semin Ophthalmol. 2015;30(5-6):364-71. doi: 10.3109/08820538.2013.874490. Epub 2014 Feb 27. PMID 24571684
- [Result] Gatinel D, Malet J, Hoang-Xuan T, Azar DT. Corneal elevation topography: best fit sphere, elevation distance, asphericity, toricity, and clinical implications. Cornea. 2011 May;30(5):508-15. doi: 10.1097/ICO.0b013e3181fb4fa7. PMID 21107250
- [Result] Kamiya K, Ishii R, Shimizu K, Igarashi A. Evaluation of corneal elevation, pachymetry and keratometry in keratoconic eyes with respect to the stage of Amsler-Krumeich classification. Br J Ophthalmol. 2014 Apr;98(4):459-63. doi: 10.1136/bjophthalmol-2013-304132. Epub 2014 Jan 23. PMID 24457362
- [Result] Kara N, Altinkaynak H, Baz O, Goker Y. Biomechanical evaluation of cornea in topographically normal relatives of patients with keratoconus. Cornea. 2013 Mar;32(3):262-6. doi: 10.1097/ICO.0b013e3182490924. PMID 22677642
- [Result] Karimian F, Aramesh S, Rabei HM, Javadi MA, Rafati N. Topographic evaluation of relatives of patients with keratoconus. Cornea. 2008 Sep;27(8):874-8. doi: 10.1097/ICO.0b013e31816f5edc. PMID 18724146
- [Result] Kawata A, Kato S, Shimizu T, Hayashi H, Hirai S, Misawa H, Takahashi R. Aberrant splicing of human Cu/Zn superoxide dismutase (SOD1) RNA transcripts. Neuroreport. 2000 Aug 21;11(12):2649-53. doi: 10.1097/00001756-200008210-00009. PMID 10976937
- [Result] Kenney MC, Chwa M, Atilano SR, Tran A, Carballo M, Saghizadeh M, Vasiliou V, Adachi W, Brown DJ. Increased levels of catalase and cathepsin V/L2 but decreased TIMP-1 in keratoconus corneas: evidence that oxidative stress plays a role in this disorder. Invest Ophthalmol Vis Sci. 2005 Mar;46(3):823-32. doi: 10.1167/iovs.04-0549. PMID 15728537
- [Result] Kim WJ, Rabinowitz YS, Meisler DM, Wilson SE. Keratocyte apoptosis associated with keratoconus. Exp Eye Res. 1999 Nov;69(5):475-81. doi: 10.1006/exer.1999.0719. PMID 10548467
- [Result] Klyce SD. Computer-assisted corneal topography. High-resolution graphic presentation and analysis of keratoscopy. Invest Ophthalmol Vis Sci. 1984 Dec;25(12):1426-35. PMID 6511226
- [Result] Klyce SD. Chasing the suspect: keratoconus. Br J Ophthalmol. 2009 Jul;93(7):845-7. doi: 10.1136/bjo.2008.147371. No abstract available. PMID 19553507
- [Result] Koenig SB, Smith RW. Keratoconus and corneal hydrops associated with compulsive eye rubbing. Refract Corneal Surg. 1993 Sep-Oct;9(5):383-4. No abstract available. PMID 8241044
- [Result] Kosker M, Suri K, Hammersmith KM, Nassef AH, Nagra PK, Rapuano CJ. Another look at the association between diabetes and keratoconus. Cornea. 2014 Aug;33(8):774-9. doi: 10.1097/ICO.0000000000000167. PMID 24915014
- [Result] Kuo IC, Broman A, Pirouzmanesh A, Melia M. Is there an association between diabetes and keratoconus? Ophthalmology. 2006 Feb;113(2):184-90. doi: 10.1016/j.ophtha.2005.10.009. Epub 2005 Dec 20. PMID 16368147
- [Result] Lechner J, Porter LF, Rice A, Vitart V, Armstrong DJ, Schorderet DF, Munier FL, Wright AF, Inglehearn CF, Black GC, Simpson DA, Manson F, Willoughby CE. Enrichment of pathogenic alleles in the brittle cornea gene, ZNF469, in keratoconus. Hum Mol Genet. 2014 Oct 15;23(20):5527-35. doi: 10.1093/hmg/ddu253. Epub 2014 Jun 3. PMID 24895405
- [Result] Lee JE, Oum BS, Choi HY, Lee SU, Lee JS. Evaluation of differentially expressed genes identified in keratoconus. Mol Vis. 2009 Nov 28;15:2480-7. PMID 19956410
- [Result] Lema I, Brea D, Rodriguez-Gonzalez R, Diez-Feijoo E, Sobrino T. Proteomic analysis of the tear film in patients with keratoconus. Mol Vis. 2010 Oct 13;16:2055-61. PMID 21042560
- [Result] Li X, Bykhovskaya Y, Haritunians T, Siscovick D, Aldave A, Szczotka-Flynn L, Iyengar SK, Rotter JI, Taylor KD, Rabinowitz YS. A genome-wide association study identifies a potential novel gene locus for keratoconus, one of the commonest causes for corneal transplantation in developed countries. Hum Mol Genet. 2012 Jan 15;21(2):421-9. doi: 10.1093/hmg/ddr460. Epub 2011 Oct 6. PMID 21979947
- [Result] Li X, Rabinowitz YS, Tang YG, Picornell Y, Taylor KD, Hu M, Yang H. Two-stage genome-wide linkage scan in keratoconus sib pair families. Invest Ophthalmol Vis Sci. 2006 Sep;47(9):3791-5. doi: 10.1167/iovs.06-0214. PMID 16936089
- [Result] Lim L, Wei RH, Chan WK, Tan DT. Evaluation of keratoconus in Asians: role of Orbscan II and Tomey TMS-2 corneal topography. Am J Ophthalmol. 2007 Mar;143(3):390-400. doi: 10.1016/j.ajo.2006.11.030. Epub 2006 Dec 21. PMID 17224118
- [Result] Liskova P, Hysi PG, Waseem N, Ebenezer ND, Bhattacharya SS, Tuft SJ. Evidence for keratoconus susceptibility locus on chromosome 14: a genome-wide linkage screen using single-nucleotide polymorphism markers. Arch Ophthalmol. 2010 Sep;128(9):1191-5. doi: 10.1001/archophthalmol.2010.200. PMID 20837804
- [Result] Balasubramanian SA, Pye DC, Willcox MD. Are proteinases the reason for keratoconus? Curr Eye Res. 2010 Mar;35(3):185-91. doi: 10.3109/02713680903477824. PMID 20373876
- [Result] Balasubramanian SA, Mohan S, Pye DC, Willcox MD. Proteases, proteolysis and inflammatory molecules in the tears of people with keratoconus. Acta Ophthalmol. 2012 Jun;90(4):e303-9. doi: 10.1111/j.1755-3768.2011.02369.x. Epub 2012 Mar 13. PMID 22413749
- [Result] Macsai MS, Varley GA, Krachmer JH. Development of keratoconus after contact lens wear. Patient characteristics. Arch Ophthalmol. 1990 Apr;108(4):534-8. doi: 10.1001/archopht.1990.01070060082054. PMID 2322155
- [Result] Saad A, Gatinel D. Evaluation of total and corneal wavefront high order aberrations for the detection of forme fruste keratoconus. Invest Ophthalmol Vis Sci. 2012 May 17;53(6):2978-92. doi: 10.1167/iovs.11-8803. PMID 22427590
- [Result] Bessho K, Maeda N, Kuroda T, Fujikado T, Tano Y, Oshika T. Automated keratoconus detection using height data of anterior and posterior corneal surfaces. Jpn J Ophthalmol. 2006 Sep-Oct;50(5):409-416. doi: 10.1007/s10384-006-0349-6. PMID 17013692
- [Result] Maeda N, Klyce SD, Smolek MK, Thompson HW. Automated keratoconus screening with corneal topography analysis. Invest Ophthalmol Vis Sci. 1994 May;35(6):2749-57. PMID 8188468
- [Result] Matthews FJ, Cook SD, Majid MA, Dick AD, Smith VA. Changes in the balance of the tissue inhibitor of matrix metalloproteinases (TIMPs)-1 and -3 may promote keratocyte apoptosis in keratoconus. Exp Eye Res. 2007 Jun;84(6):1125-34. doi: 10.1016/j.exer.2007.02.013. Epub 2007 Mar 7. PMID 17449031
- [Result] McGhee CN. 2008 Sir Norman McAlister Gregg Lecture: 150 years of practical observations on the conical cornea--what have we learned? Clin Exp Ophthalmol. 2009 Mar;37(2):160-76. doi: 10.1111/j.1442-9071.2009.02009.x. PMID 19426404
- [Result] Mikami T, Meguro A, Teshigawara T, Takeuchi M, Uemoto R, Kawagoe T, Nomura E, Asukata Y, Ishioka M, Iwasaki M, Fukagawa K, Konomi K, Shimazaki J, Nishida T, Mizuki N. Interleukin 1 beta promoter polymorphism is associated with keratoconus in a Japanese population. Mol Vis. 2013 Apr 11;19:845-51. Print 2013. PMID 23592922
- [Result] Nielsen K, Hjortdal J, Pihlmann M, Corydon TJ. Update on the keratoconus genetics. Acta Ophthalmol. 2013 Mar;91(2):106-13. doi: 10.1111/j.1755-3768.2012.02400.x. Epub 2012 Apr 4. PMID 22471291
- [Result] Chan S, Freund PR, MacDonald I. Advances in the genetics of eye diseases. Curr Opin Pediatr. 2013 Dec;25(6):645-52. doi: 10.1097/MOP.0000000000000026. PMID 24126856
- [Result] Nilforoushan MR, Speaker M, Marmor M, Abramson J, Tullo W, Morschauser D, Latkany R. Comparative evaluation of refractive surgery candidates with Placido topography, Orbscan II, Pentacam, and wavefront analysis. J Cataract Refract Surg. 2008 Apr;34(4):623-31. doi: 10.1016/j.jcrs.2007.11.054. PMID 18361985
- [Result] Ohtoshi A, Wang SW, Maeda H, Saszik SM, Frishman LJ, Klein WH, Behringer RR. Regulation of retinal cone bipolar cell differentiation and photopic vision by the CVC homeobox gene Vsx1. Curr Biol. 2004 Mar 23;14(6):530-6. doi: 10.1016/j.cub.2004.02.027. PMID 15043821
- [Result] Ortak H, Sogut E, Tas U, Mesci C, Mendil D. The relation between keratoconus and plasma levels of MMP-2, zinc, and SOD. Cornea. 2012 Sep;31(9):1048-51. doi: 10.1097/ICO.0b013e318254c028. PMID 22580443
- [Result] Owens H, Gamble GD, Bjornholdt MC, Boyce NK, Keung L. Topographic indications of emerging keratoconus in teenage New Zealanders. Cornea. 2007 Apr;26(3):312-8. doi: 10.1097/ICO.0b013e31802f8d87. PMID 17413959
- [Result] Pihlblad MS, Schaefer DP. Eyelid laxity, obesity, and obstructive sleep apnea in keratoconus. Cornea. 2013 Sep;32(9):1232-6. doi: 10.1097/ICO.0b013e318281e755. PMID 23471083
- [Result] Parker JS, van Dijk K, Melles GR. Treatment options for advanced keratoconus: A review. Surv Ophthalmol. 2015 Sep-Oct;60(5):459-80. doi: 10.1016/j.survophthal.2015.02.004. Epub 2015 Mar 5. PMID 26077628
- [Result] Randleman JB, Dupps WJ Jr, Santhiago MR, Rabinowitz YS, Koch DD, Stulting RD, Klyce SD. Screening for Keratoconus and Related Ectatic Corneal Disorders. Cornea. 2015 Aug;34(8):e20-2. doi: 10.1097/ICO.0000000000000500. No abstract available. PMID 26075463
- [Result] Steinberg J, Aubke-Schultz S, Frings A, Hulle J, Druchkiv V, Richard G, Katz T, Linke SJ. Correlation of the KISA% index and Scheimpflug tomography in 'normal', 'subclinical', 'keratoconus-suspect' and 'clinically manifest' keratoconus eyes. Acta Ophthalmol. 2015 May;93(3):e199-207. doi: 10.1111/aos.12590. PMID 25873278
- [Result] Tang YG, Picornell Y, Su X, Li X, Yang H, Rabinowitz YS. Three VSX1 gene mutations, L159M, R166W, and H244R, are not associated with keratoconus. Cornea. 2008 Feb;27(2):189-92. doi: 10.1097/ICO.0b013e31815a50e7. PMID 18216574
- [Result] Rabinowitz YS. The genetics of keratoconus. Ophthalmol Clin North Am. 2003 Dec;16(4):607-20, vii. doi: 10.1016/s0896-1549(03)00099-3. PMID 14741001
- [Result] Wang Y, Rabinowitz YS, Rotter JI, Yang H. Genetic epidemiological study of keratoconus: evidence for major gene determination. Am J Med Genet. 2000 Aug 28;93(5):403-9. PMID 10951465
- [Result] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Result] Romero-Jimenez M, Santodomingo-Rubido J, Wolffsohn JS. Keratoconus: a review. Cont Lens Anterior Eye. 2010 Aug;33(4):157-66; quiz 205. doi: 10.1016/j.clae.2010.04.006. PMID 20537579
- [Result] Rose NJ, Mackay K, Byers PH, Dalgleish R. A Gly238Ser substitution in the alpha 2 chain of type I collagen results in osteogenesis imperfecta type III. Hum Genet. 1995 Feb;95(2):215-8. doi: 10.1007/BF00209405. PMID 7860070
- [Result] Saee-Rad S, Raoofian R, Mahbod M, Miraftab M, Mojarrad M, Asgari S, Rezvan F, Hashemi H. Analysis of superoxide dismutase 1, dual-specificity phosphatase 1, and transforming growth factor, beta 1 genes expression in keratoconic and non-keratoconic corneas. Mol Vis. 2013 Dec 8;19:2501-7. eCollection 2013. PMID 24339725
- [Result] Saee-Rad S, Hashemi H, Miraftab M, Noori-Daloii MR, Chaleshtori MH, Raoofian R, Jafari F, Greene W, Fakhraie G, Rezvan F, Heidari M. Mutation analysis of VSX1 and SOD1 in Iranian patients with keratoconus. Mol Vis. 2011;17:3128-36. Epub 2011 Nov 30. PMID 22171159
- [Result] Semina EV, Mintz-Hittner HA, Murray JC. Isolation and characterization of a novel human paired-like homeodomain-containing transcription factor gene, VSX1, expressed in ocular tissues. Genomics. 2000 Jan 15;63(2):289-93. doi: 10.1006/geno.1999.6093. PMID 10673340
- [Result] Sherwin T, Brookes NH. Morphological changes in keratoconus: pathology or pathogenesis. Clin Exp Ophthalmol. 2004 Apr;32(2):211-7. doi: 10.1111/j.1442-9071.2004.00805.x. PMID 15068441
- [Result] Spoerl E, Raiskup-Wolf F, Kuhlisch E, Pillunat LE. Cigarette smoking is negatively associated with keratoconus. J Refract Surg. 2008 Sep;24(7):S737-40. doi: 10.3928/1081597X-20080901-18. PMID 18811121
- [Result] Stabuc-Silih M, Strazisar M, Hawlina M, Glavac D. Absence of pathogenic mutations in VSX1 and SOD1 genes in patients with keratoconus. Cornea. 2010 Feb;29(2):172-6. doi: 10.1097/ICO.0b013e3181aebf7a. PMID 20023586
- [Result] Swartz T, Marten L, Wang M. Measuring the cornea: the latest developments in corneal topography. Curr Opin Ophthalmol. 2007 Jul;18(4):325-33. doi: 10.1097/ICU.0b013e3281ca7121. PMID 17568210
- [Result] Tai LY, Khaw KW, Ng CM, Subrayan V. Central corneal thickness measurements with different imaging devices and ultrasound pachymetry. Cornea. 2013 Jun;32(6):766-71. doi: 10.1097/ICO.0b013e318269938d. PMID 23095499
- [Result] Tuft SJ, Hassan H, George S, Frazer DG, Willoughby CE, Liskova P. Keratoconus in 18 pairs of twins. Acta Ophthalmol. 2012 Sep;90(6):e482-6. doi: 10.1111/j.1755-3768.2012.02448.x. Epub 2012 Jun 8. PMID 22682160
- [Result] Ucakhan OO, Cetinkor V, Ozkan M, Kanpolat A. Evaluation of Scheimpflug imaging parameters in subclinical keratoconus, keratoconus, and normal eyes. J Cataract Refract Surg. 2011 Jun;37(6):1116-24. doi: 10.1016/j.jcrs.2010.12.049. PMID 21596255
- [Result] Udar N, Atilano SR, Brown DJ, Holguin B, Small K, Nesburn AB, Kenney MC. SOD1: a candidate gene for keratoconus. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3345-51. doi: 10.1167/iovs.05-1500. PMID 16877401
- [Result] Vazirani J, Basu S. Keratoconus: current perspectives. Clin Ophthalmol. 2013;7:2019-30. doi: 10.2147/OPTH.S50119. Epub 2013 Oct 14. PMID 24143069
- [Result] Wagner H, Barr JT, Zadnik K. Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study: methods and findings to date. Cont Lens Anterior Eye. 2007 Sep;30(4):223-32. doi: 10.1016/j.clae.2007.03.001. Epub 2007 May 3. PMID 17481941
- [Result] Wegener A, Laser-Junga H. Photography of the anterior eye segment according to Scheimpflug's principle: options and limitations - a review. Clin Exp Ophthalmol. 2009 Jan;37(1):144-54. doi: 10.1111/j.1442-9071.2009.02018.x. PMID 19338611
- [Result] Weissman BA, Ehrlich M, Levenson JE, Pettit TH. Four cases of keratoconus and posterior polymorphous corneal dystrophy. Optom Vis Sci. 1989 Apr;66(4):243-6. doi: 10.1097/00006324-198904000-00012. PMID 2786175
- [Result] Wilson SE, He YG, Weng J, Li Q, McDowall AW, Vital M, Chwang EL. Epithelial injury induces keratocyte apoptosis: hypothesized role for the interleukin-1 system in the modulation of corneal tissue organization and wound healing. Exp Eye Res. 1996 Apr;62(4):325-7. doi: 10.1006/exer.1996.0038. PMID 8795451
- [Result] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Result] Wojcik KA, Blasiak J, Szaflik J, Szaflik JP. Role of biochemical factors in the pathogenesis of keratoconus. Acta Biochim Pol. 2014;61(1):55-62. Epub 2014 Mar 18. PMID 24644548
- [Result] Zadnik K, Barr JT, Edrington TB, Everett DF, Jameson M, McMahon TT, Shin JA, Sterling JL, Wagner H, Gordon MO. Baseline findings in the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study. Invest Ophthalmol Vis Sci. 1998 Dec;39(13):2537-46. PMID 9856763
- [Result] Zelko IN, Mariani TJ, Folz RJ. Superoxide dismutase multigene family: a comparison of the CuZn-SOD (SOD1), Mn-SOD (SOD2), and EC-SOD (SOD3) gene structures, evolution, and expression. Free Radic Biol Med. 2002 Aug 1;33(3):337-49. doi: 10.1016/s0891-5849(02)00905-x. PMID 12126755